CLINICAL TRIAL: NCT02276885
Title: Prone Partial Breast Irradiation (PBI): A Prospective Randomized Trial Comparing Five Versus Three Fractions
Brief Title: Prone Partial Breast Irradiation (PBI): a Prospective Randomized Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-01306
Record Dates: First submitted 2014-10-24; First posted 2014-10-28 (Estimated); Results first posted 2024-12-31 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: breast; cancer; breast cancer; prone; partial breast irradiation; PBI
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PBI Radiotherapy 6 Gy (Experimental): Prone partial breast irradiation of 6 Gy x 5 over 5 days, on five consecutive days
  Interventions: Radiation: PBI Radiotherapy 6 Gy
- PBI Radiotherapy 8 Gy (Experimental): Prone partial breast irradiation of 8 Gy x 3 over 5 days, every other day
  Interventions: Radiation: PBI Radiotherapy 8 Gy

INTERVENTIONS:
Radiation: PBI Radiotherapy 6 Gy — Patients will receive 3D-Conformal or Intensity Modulated Radiation Therapy (IMRT) of 6 Gy x 5, over 5 consecutive days
  Other Names: 3D-Conformal; Intensity Modulated Radiation Therapy; Prone partial breast irradiation
  Arms: PBI Radiotherapy 6 Gy
Radiation: PBI Radiotherapy 8 Gy — Patients will receive 3D-Conformal or Intensity Modulated Radiation Therapy (IMRT) of 8 Gy x 3, over 5 days, every other day
  Other Names: 3D-Conformal; Intensity Modulated Radiation Therapy; Prone partial breast irradiation
  Arms: PBI Radiotherapy 8 Gy

SUMMARY:
The purpose of this study is to test whether a radiotherapy regimen of 8 GY x 3 days over 5 days (every other day) is as safe (well-tolerated) and effective as 6 Gy x 5 over five consecutive days

DETAILED DESCRIPTION:
Despite the fact that less extensive experience than that of brachytherapy is available, PBI delivery through an external-beam has many advantages. First of all, it is likely to be more acceptable to the patient since it is non-invasive and it does not require a surgical procedure or anesthesia. Moreover, since it is delivered after surgery, the pathological analysis of the segmental mastectomy specimen is available to inform the selection of the best candidates. In addition, EB-PBI is likely to become more widely reproducible, since it does not rely on the experience and skills of the radiation oncologist performing the brachytherapy implant. Besides, once the technique is established, it can be widely applied at any facility provided with a linear accelerator, without the risk presented by some brachytherapy approaches that can not be completed because of the unfavorable interplay of patient's anatomy with the technical limitations of the applicator.

The women in this study will receive either 5 or 3 radiation fractions to the tumor bed. We have chosen to study T1 post menopausal women because in this subset: 1) the tumor is small enough to be treated by partial breast radiation 2) the odds of having multicentric disease are low, making it ethical to avoid whole breast irradiation, 3) the most benefit from reducing the radiation schedule from 5 to 3 could be expected.

All patients will receive either 8 Gy x 3 over 5 days, every other day or 6 Gy x 5 over 5 days, on five consecutive days

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women defined as either:

  1. at least 2 years without menstrual period
  2. patients older than 50 with serological evidence of post-menopausal status
  3. hysterectomized patients of any age with FSH confirmation of post- menopausal status
* pT1 breast cancer, excised with negative margins. Criteria for low risk-pTis:

  1. Screen-detected
  2. Low to intermediate nuclear grade
  3. < 2.5cm in size
  4. Resected with negative margins at >3mm)
* clinically N0 or pN0 or sentinel node negative breast cancer

Exclusion Criteria:

* previous radiation therapy to the ipsilateral breast
* presence of a proportion of DCIS in the core biopsy specimen which is compatible with extensive intraductal component (EIC)

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2026-12-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Naamit Gerber, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PBI Radiotherapy 6 Gy | PBI Radiotherapy 8 Gy
Started | 144 | 140
Completed | 137 | 138
Not Completed | 7 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 5 | 2

BASELINE CHARACTERISTICS:
Population: Baseline data was collected and analyzed for all participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | PBI Radiotherapy 6 Gy | PBI Radiotherapy 8 Gy | Total
Number analyzed (Participants) | 144 | 140 | 284
Age, Continuous [Mean (Full Range); unit: years] | 69 [51 to 85] | 68 [48 to 87] | 68 [48 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 140 | 284
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 9 | 22
  Not Hispanic or Latino | 123 | 123 | 246
  Unknown or Not Reported | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 4 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 9 | 19
  White | 110 | 109 | 219
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 18 | 33
Region of Enrollment [Number; unit: participants]
  United States | 144 | 140 | 284

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade 2 or 3 Fibrosis
Time Frame: 60 months
Measure: Number; unit: percentage of participants
Arm/Group | PBI Radiotherapy 6 Gy | PBI Radiotherapy 8 Gy
Number analyzed (Participants) | 137 | 138
percentage of participants | 18.30 | 12.30

2. Secondary Outcome: Rate of Isolated Local/Regional Recurrences
Time Frame: 1 year post randomization
Reporting Status: Not Posted, anticipated posting 2027-12

3. Secondary Outcome: Rate of Concomitant Local/Regional and Distant Recurrences
Time Frame: 1 year post randomization
Reporting Status: Not Posted, anticipated posting 2027-12

4. Secondary Outcome: Rate of Isolated Local/Regional Recurrences
Time Frame: 2 years post randomization
Reporting Status: Not Posted, anticipated posting 2027-12

5. Secondary Outcome: Rate of Concomitant Local/Regional and Distant Recurrences
Time Frame: 2 years post randomization
Reporting Status: Not Posted, anticipated posting 2027-12

6. Secondary Outcome: Rate of Isolated Local/Regional Recurrences
Time Frame: 3 years post randomization
Reporting Status: Not Posted, anticipated posting 2027-12

7. Secondary Outcome: Rate of Concomitant Local/Regional and Distant Recurrences
Time Frame: 3 years post randomization
Reporting Status: Not Posted, anticipated posting 2027-12

ADVERSE EVENTS:
Time Frame: From the date that subjects signed the ICF until the 5 years follow up visit (EOS)
Description: Clinical assessment
Arm/Group | PBI Radiotherapy 6 Gy | PBI Radiotherapy 8 Gy
All-Cause Mortality (participants affected / at risk) | 4/144 | 4/140
Serious Adverse Events (participants affected / at risk) | 0/144 | 1/140
Other Adverse Events (participants affected / at risk) | 144/144 | 140/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PBI Radiotherapy 6 Gy (N=144) | PBI Radiotherapy 8 Gy (N=140)
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PBI Radiotherapy 6 Gy (N=144) | PBI Radiotherapy 8 Gy (N=140)
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Agitation (Psychiatric disorders) | 1 | 2
Allergic reaction (Immune system disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 4
Amnesia (Nervous system disorders) | 1 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 3
Anxiety (Psychiatric disorders) | 5 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 39 | 35
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Breast Asymmetry (Musculoskeletal and connective tissue disorders) | 18 | 15
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 11
Bloating (Gastrointestinal disorders) | 2 | 0
Myelodysplastic syndrome (Blood and lymphatic system disorders) | 1 | 0
Cervical Adenopathy (Blood and lymphatic system disorders) | 1 | 0
Body odor (Skin and subcutaneous tissue disorders) | 0 | 1
Breast Atrophy (Reproductive system and breast disorders) | 36 | 41
Brain dx other - fogsy (Nervous system disorders) | 0 | 1
Breast disorder: tingling (Reproductive system and breast disorders) | 0 | 2
Breast disorder: twinges (Reproductive system and breast disorders) | 0 | 1
Breast infection (Infections and infestations) | 2 | 0
Breast pain (Reproductive system and breast disorders) | 36 | 25
Bruising (Injury, poisoning and procedural complications) | 1 | 2
Palpitations (Cardiac disorders) | 3 | 3
Left coronary artery artherosclerotic dx (Cardiac disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 2 | 1
Breast retraction (Reproductive system and breast disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 7 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1
Concentration impairment (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Cushingoid (Endocrine disorders) | 1 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 101 | 82
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 1
Weight Loss (Investigations) | 3 | 2
Depression (Psychiatric disorders) | 2 | 7
Weight Gain (Investigations) | 8 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Watering eyes (Eye disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 4 | 3
Dizziness (Nervous system disorders) | 3 | 5
Vomiting (Gastrointestinal disorders) | 3 | 1
Urinary Tract Infection (Infections and infestations) | 3 | 4
Discomfort from table positioning (Investigations) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 11
Urinary Incontinence (Renal and urinary disorders) | 5 | 0
Upper respiratory infection (Infections and infestations) | 7 | 3
Urinary Frequency (Renal and urinary disorders) | 2 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 1 | 0
Vaginal Dryness (Reproductive system and breast disorders) | 0 | 3
Vaginal Hemorrhage (Reproductive system and breast disorders) | 0 | 1
Superficial Soft TIssue Fibrosis (Musculoskeletal and connective tissue disorders) | 49 | 45
Skin induration (Skin and subcutaneous tissue disorders) | 9 | 4
skin infection (Infections and infestations) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 12 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Edema limbs (General disorders) | 2 | 2
Elevated IgE (Immune system disorders) | 0 | 1
Hypercholesteremia (Endocrine disorders) | 1 | 0
Diabetes (Endocrine disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Esophageal ulcer (Gastrointestinal disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 6 | 3
Wound infection (Infections and infestations) | 1 | 0
Redness (Eye disorders) | 3 | 1
Fall (Injury, poisoning and procedural complications) | 7 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 4
Fatigue (General disorders) | 110 | 122
Nausea (Gastrointestinal disorders) | 9 | 5
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 | 9
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 | 8
Fever (General disorders) | 0 | 2
Flu like symptoms (General disorders) | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 4 | 3
Paresthesia (Nervous system disorders) | 2 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gait disturbance (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Abdominal Cramping (Gastrointestinal disorders) | 1 | 0
GI Symptoms (Gastrointestinal disorders) | 0 | 1
Diverticulosis (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 9
telangiectasia (Skin and subcutaneous tissue disorders) | 6 | 1
syncope (Nervous system disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 1
nipple deformity (Reproductive system and breast disorders) | 2 | 2
non-cardiac chest pain (General disorders) | 1 | 2
stomach pain (Gastrointestinal disorders) | 1 | 1
Papulopustular rash (Infections and infestations) | 2 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 4
joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 3 | 5
lymphedema (Vascular disorders) | 9 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 1
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 5 | 3
Peripheral motor neuropathy (Nervous system disorders) | 0 | 3
periorbital edema (Eye disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 | 15
Hypertension (Vascular disorders) | 1 | 2
Hematuria (Renal and urinary disorders) | 1 | 2
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 78 | 67
Hot Flashes (Vascular disorders) | 64 | 67
Pain (General disorders) | 46 | 43
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Heart failure (Cardiac disorders) | 1 | 0
Hematoma (Vascular disorders) | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Skin Induration (Skin and subcutaneous tissue disorders) | 2 | 0
Giardia (Infections and infestations) | 0 | 1
Elevated AFP (Hepatobiliary disorders) | 1 | 0
Hepatobiliary dx - Other: hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Hepatobiliary dx- Other: LFTs/increased/transiminitis (Hepatobiliary disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Cellulitis (Skin Infection) (Infections and infestations) | 2 | 1
Osteomyelitis (Infections and infestations) | 1 | 1
COVID 19 (Infections and infestations) | 1 | 1
localized edema (General disorders) | 28 | 26
Lyme disease (Infections and infestations) | 0 | 1
Pelvic prolapse (Injury, poisoning and procedural complications) | 1 | 0
Right Inguinal Hernia (Injury, poisoning and procedural complications) | 0 | 1
Knee sprain (Injury, poisoning and procedural complications) | 0 | 1
Arm/Wrist Broken (Injury, poisoning and procedural complications) | 1 | 0
L4-L5 Central and Lateral Stenosis (Injury, poisoning and procedural complications) | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 2 | 3
Irregular heart rhythm (Cardiac disorders) | 0 | 1
Irritability (Psychiatric disorders) | 1 | 0
Breast abscess (Reproductive system and breast disorders) | 1 | 1
Breast dimpling (Reproductive system and breast disorders) | 7 | 7
Pruritis (Skin and subcutaneous tissue disorders) | 30 | 30
Breast skin thickening (Reproductive system and breast disorders) | 8 | 6
Breast seborrheic keratosis (Reproductive system and breast disorders) | 1 | 2
Eye infection (Infections and infestations) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 2
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Arm Tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Carpal Tunnel (Musculoskeletal and connective tissue disorders) | 1 | 2
Hemiparesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Shoulder) (Musculoskeletal and connective tissue disorders) | 1 | 0
Arm pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Knee pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Leg Cramps (Musculoskeletal and connective tissue disorders) | 0 | 1
Hand stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
LE Stiffness Intermittent (Musculoskeletal and connective tissue disorders) | 0 | 1
Tissue Defect LLIQ with Arm Elevation (Musculoskeletal and connective tissue disorders) | 1 | 0
Radiculitis (Nervous system disorders) | 1 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Degenerative joint desease (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Alzheimer (Nervous system disorders) | 0 | 2
Imbalance (Nervous system disorders) | 1 | 0
Aversion to Certain Foods (Nervous system disorders) | 1 | 0
Personage turner syndrome (Nervous system disorders) | 1 | 0
Mental Fogginess (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Right Elbow Ulnar Nerve Entrapment (Nervous system disorders) | 0 | 1
Meningioma (Nervous system disorders) | 0 | 1
Balancing Issues (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
amyloid angiopathy (Nervous system disorders) | 1 | 0
erythrodysesthesia syndrome (Nervous system disorders) | 0 | 1
Mood changes (Psychiatric disorders) | 1 | 0
Vasovagal reaction (Nervous system disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cold flashes (Vascular disorders) | 0 | 1
Breast intertrigo candida (Reproductive system and breast disorders) | 2 | 2
Breast Surgical Incision Drainage (Surgical and medical procedures) | 1 | 0
Breast burning sensation (Skin and subcutaneous tissue disorders) | 1 | 4
Papillary Urethelial Carcinoma (Renal and urinary disorders) | 0 | 1
Intermittent increased urinary frequency post BCG treatment (Renal and urinary disorders) | 1 | 0
vaginal spotting (Reproductive system and breast disorders) | 1 | 0
vaginal atrophy (Reproductive system and breast disorders) | 1 | 0
Ovarian Mass/Fibroma (Reproductive system and breast disorders) | 1 | 0
Nipple Discharge (Reproductive system and breast disorders) | 0 | 2
Breast red/blue discoloration (Reproductive system and breast disorders) | 0 | 1
Vaginal Bleeding (Reproductive system and breast disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Aortic Thrombosis (Cardiac disorders) | 0 | 1
breast swelling (Reproductive system and breast disorders) | 1 | 1
uterine fibroid (Reproductive system and breast disorders) | 1 | 0
breast sx site hypersensation (Reproductive system and breast disorders) | 0 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Contact dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Difficult Coping With Diagnosis (Psychiatric disorders) | 1 | 0
Fibrocystic changes (Reproductive system and breast disorders) | 1 | 0
shoulder discomfort due to positioning (Musculoskeletal and connective tissue disorders) | 0 | 1
LLQ of Left Breast (Skin and subcutaneous tissue disorders) | 1 | 0
Scar tissueat sx site (Skin and subcutaneous tissue disorders) | 3 | 1
Skin breakdown (breast) (Skin and subcutaneous tissue disorders) | 3 | 0
Pre-ulcerative Calluses Feet (Skin and subcutaneous tissue disorders) | 0 | 1
Hemangioma Right Hepatic (Hepatobiliary disorders) | 1 | 0
Breast Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Breast Skin Reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Breast LUQ Tissue Defect (Reproductive system and breast disorders) | 1 | 2
Lip sore (Skin and subcutaneous tissue disorders) | 1 | 0
Facial Redness (Skin and subcutaneous tissue disorders) | 1 | 0
fat necrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Mouth Swelling (Skin and subcutaneous tissue disorders) | 1 | 0
Contraction at Surgical Site (braest) (Reproductive system and breast disorders) | 1 | 0
Papule/Folliculitis Breast Fold (Skin and subcutaneous tissue disorders) | 1 | 0
Neck Nodule (Skin and subcutaneous tissue disorders) | 1 | 0
Breast incision surgical defect (Reproductive system and breast disorders) | 1 | 0
chest wall nodule (Skin and subcutaneous tissue disorders) | 1 | 0
LIQ Breast Mass (Reproductive system and breast disorders) | 0 | 1
Pre-cancerous Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Hand rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders: other - Tick bite (Skin and subcutaneous tissue disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Vaginal pain (Reproductive system and breast disorders) | 0 | 1
Ground glass opacity (GGO) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other: Axilla pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other: Keloid (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other: Adhesive capsulitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Blurred vision (Eye disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT02276885/Prot_SAP_000.pdf